CLINICAL TRIAL: NCT00484562
Title: A Randomized, Multi-arm Repeated Measures Prospective Study Comparing Different Modalities of Portable Oxygen Delivery During Assessment of Functional Exercise Capacity
Brief Title: Prospective Study Comparing Different Modalities of Oxygen Delivery During Assessment of Functional Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060507
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: COPD
Keywords: oxygen; COPD; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard oxygen delivery system (Active Comparator): Standard oxygen tank with pulse dose regulator
  Interventions: Device: Standard oxygen delivery system
- Homefill oxygen delivery system (Active Comparator): Homefill oxygen delivery system, pre-filled from a larger oxygen concentrator base unit.
  Interventions: Device: Homefill oxygen delivery system
- Helios oxygen delivery system (Active Comparator): Liquid oxygen portable system pre-filled from a larger liquid oxygen tank
  Interventions: Device: Helios oxygen delivery system
- FreeStyle oxygen system (Active Comparator): portable battery-powered oxygen concentrator delivery system
  Interventions: Device: FreeStyle oxygen system

INTERVENTIONS:
Device: Standard oxygen delivery system — Standard oxygen tank with pulse dose regulator
  Arms: Standard oxygen delivery system
Device: Homefill oxygen delivery system — Homefill oxygen delivery system, pre-filled from a larger oxygen concentrator base unit.
  Arms: Homefill oxygen delivery system
Device: Helios oxygen delivery system — Liquid oxygen portable system pre-filled from a larger liquid oxygen tank
  Arms: Helios oxygen delivery system
Device: FreeStyle oxygen system — portable battery-powered oxygen concentrator delivery system
  Arms: FreeStyle oxygen system

SUMMARY:
Objectives:

The objective of this study is to determine if any differences exist between the varying modes of portable oxygen delivery systems including liquid oxygen, a portable concentrator, portable devices filled at home from a concentrator, and medical grade compressed oxygen (either an M6 size or D size cylinder).

Hypothesis:

Patients who are prescribed LTOT will show similar physiologic responses to exercise when using differing modalities of portable oxygen delivery systems.

DETAILED DESCRIPTION:
There are over 900,000 individuals currently utilizing Long Term Oxygen Therapy (LTOT) in this country. LTOT is administered by using one or a combination of three basic delivery systems: compressed gas cylinder, liquid oxygen system, and oxygen concentrator. Each of the base oxygen delivery systems has unique advantages and disadvantages regarding operation, function, and cost.

The majority of LTOT users require oxygen during ambulation. Within the home this is accomplished by a 20-50-foot extension tubing. Extending the length of the tubing allows the user (patient) to ambulate up to the extended distance from the base oxygen delivery system. Limitations are of course, the distance, becoming entangled in the tubing and it is not conducive for short trips such as to the mailbox.

Ambulation outside the home, however, requires the use of a "portable oxygen system". Put simplistically, portable oxygen systems are miniaturized versions of the base systems. Here also, each particular delivery system has inherent advantages and disadvantages.

An important development in portable oxygen systems has been the advent of pulse-dose technology. Pulse-dose technology allows both the gaseous and liquid portable systems to conserve oxygen delivery. During the inspiratory phase of breathing a solenoid control valve opens "dosing" a bolus of gas flow through the cannula. Unlike traditional continuous-flow cannula, where oxygen is delivered during both the inspiratory and expiratory cycle, pulse-dose technology only delivers oxygen during in an inspiratory phase of breathing. Oxygen flow that is delivered only during inspiration results in less total oxygen consumption. This in-turn allows relatively small portable oxygen systems to be more efficient and last longer. Such efficiency is not only important to the patient, but also to the Home Medical Equipment (HME) provider. Portable oxygen systems that incorporate pulse-dose technology typically decrease the home visits required to deliver to replenish the patient's oxygen supply.

One portable technology allows the patient to refill small oxygen devices in their home, but uses electricity (battery or AC) for functionality, providing economic hardship for some patients who are prescribed LTOT. Another portable technology is an actual portable oxygen concentrator that is lightweight and operates on electricity as well.

By comparison, the oxygen delivered to patients by HME providers, in either cylinder or liquid form, is an indirect product of liquefaction of air. Stringent FDA repackaging production and transfilling processes must be met. Strength and purity testing requires such "medical grade" oxygen be at least 99.5% pure. Such medical grade oxygen containers typically result in 100% oxygen being provided to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age and older)
* Current users of prescribed LTOT
* Patients who meet the Category IV classification (Very Severe) of the Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* Medicare criteria for long-term oxygen therapy (LTOT)
* Exhibit dyspnea on exertion while breathing room air
* No exacerbation of COPD within previous 6 weeks, a resting oxygen saturation of less than 90% on room air (no supplemental oxygen) and receiving LTOT with a pulse-dose generator as prescribed by a physician

Exclusion Criteria:

* Children (persons under age 18), fetuses, neonates, pregnant women, prisoners
* Unstable angina during the previous month
* Myocardial infarction during the previous month
* Resting heart rate of > 120
* Systolic blood pressure of >180mmHg
* Diastolic blood pressure of >100 mmHg
* Physical limitations which render the participant unable to walk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Determination of ability to maintain adequate oxygenation | course of study: 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shawna L Strickland, MEd, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Harry S Truman Veterans Administration Medical Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No